CLINICAL TRIAL: NCT04764565
Title: Impact of Nuun Instant on Hydration Status in Active Men and Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Memphis (Other)
Collaborators: Nuun & Company (Unknown)
Responsible Party: Principal Investigator, Richard Bloomer, Dean of the College of Health Sciences, University of Memphis
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: PRO-FY2021-96
Record Dates: First submitted 2021-02-18; First posted 2021-02-21 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Hydration
Keywords: electrolyte; sport drink; beverage hydration index
MeSH Terms: interventions — Water

STUDY DESIGN:
Intervention Model Description: single-blind crossover
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Nuun Instant (Experimental): 2 servings of Nuun instant in 1 liter water
  Interventions: Dietary Supplement: Nuun Instant; Other: Water
- Control (Placebo Comparator): 1 liter of water
  Interventions: Other: Water
- Nuun Electrolyte (Experimental): 2.1 servings of Nuun Electrolyte in 1 liter water
  Interventions: Other: Water; Dietary Supplement: Nuun Electrolyte

INTERVENTIONS:
Dietary Supplement: Nuun Instant — Contains (per 11 gram serving) the following: 7 grams of carbohydrate, calcium (20mg, 2%DV), sodium (520mg, 23%DV), potassium (385mg, 8%DV), magnesium (8mg, 2%DV), chloride (250mg, 10%DV), and 100% of vitamin C (90mg) and B12 (2.4 mcg).
  Arms: Nuun Instant
Other: Water — water
Dietary Supplement: Nuun Electrolyte — Citric Acid, Dextrose, Sodium Bicarbonate, Potassium Bicarbonate, Sodium Carbonate, Natural Flavors, Potassium Chloride, Malic Acid, Magnesium Carbonate, Calcium Carbonate, Stevia Leaf Extract, Beet Powder Color, Safflower Oil. Nuun electrolytes contains (per tablet) the following: 3 grams of carbohydrate, calcium (15 mg, 1%DV), sodium (200 mg, 9%DV), potassium (125mg, 3%DV), magnesium (15mg, 4%DV), and chloride (75mg, 3%DV).
  Arms: Nuun Electrolyte

SUMMARY:
While Nuun Instant is commercially available and has received positive reviews from athletes, there have been no studies to date to evaluate the impact of this product on hydration status. Therefore, the purpose of this study is to determine the impact of Nuun Instant powder and new product under development called Nuun Electrolyte on hydration status in young and active men and women. We will follow a similar approach as used by Maughan and colleagues (2016) to measure the fluid balance (the difference between the amount of water consumed and passed as urine) and beverage hydration index (the relative amount of urine passed after consumption of a drink compared to water), while also measuring plasma volume using the method of Dill and Costill (1974).

DETAILED DESCRIPTION:
Maintaining adequate hydration is essential to optimal health and athletic performance. When individuals exercise (in particular in a warm environment), they can lose excessive amounts of fluids through sweating, along with necessary electrolytes (e.g., sodium, potassium, chloride). With dehydration, individuals may feel sluggish and can experience impaired physical performance.

Many attempts have been made to improve and measure the hydration status of active individuals. This typically involves the ingestion of fluids leading up to activity (typically plain water), as well as the ingestion of fluids during the activity itself (water, along with a diluted carbohydrate/electrolyte beverage). This approach seems to work well; however, some debate remains over what the best fluid is to consume, in particular related to the macronutrient type and the specific electrolyte mix.

Related to the above, it is well-accepted that electrolyte replenishment is of importance, both during and following exercise-to aid in rehydration for subsequent bouts. Electrolytes (sodium in particular) have been used for decades to aid athlete hydration and this has led to the development of various sport drinks-which also include small amounts of carbohydrate (e.g., Gatorade, Powerade). However, one problem with moderate to high carbohydrate ingestion is that some individuals experience gastrointestinal (GI) upset following carbohydrate ingestion before and during an event, despite very good physical performance outcomes. Due to this GI upset, some individuals (in particular recreationally active individuals who are not competing at high levels) rely on water alone or a very low concentrated carbohydrate beverage, and seek a method to ingest the lost electrolytes as well.

The solution to the above issues for many athletes is the use of powder "stick packs" that can be carried in bags and pockets, and simply dumped into a water bottle when needed, shaken, and consumed. They are easy to transport and provide the needed carbohydrate, as well as electrolytes to replace those that are lost through intense and/or long duration exercise.

We recently completed a study of Nuun electrolyte tablets, which provide 2 grams of carbohydrate per serving and a combination of electrolytes, provided at a relatively low percentage of the Daily Value (DV). The DV tells us how much a particular nutrient in a serving of a food product contributes to a daily diet, based on a standard 2000 calorie diet. Nuun tablets contain: calcium (13mg, 1%DV), sodium (300mg, 13%DV), potassium (150mg, 3%DV), magnesium (25mg, 6%DV), and chloride (40mg, 2%DV). Our results indicated improved hydration (based on urine output and the calculated hydration index) when subjects consumed the Nuun tablets mixed into 1 liter of water, as compared to water alone.

Nuun Instant is a new product that is similar to the Nuun tablets, but is formulated for those who may experience a significant electrolyte loss and is higher in carbohydrate as well. Specifically, the Nuun Instant product contains (per 11 gram serving) the following: 7 grams of carbohydrate, calcium (20mg, 2%DV), sodium (520mg, 23%DV), potassium (385mg, 8%DV), magnesium (8mg, 2%DV), chloride (250mg, 10%DV), and 100% of vitamin C (90mg) and B12 (2.4 mcg).

Nuun Electrolytes is a new product in development that is similar to the Nuun tablets, but with an adjusted formula. Nuun Electrolytes consist of Citric Acid, Dextrose, Sodium Bicarbonate, Potassium Bicarbonate, Sodium Carbonate, Natural Flavors, Potassium Chloride, Malic Acid, Magnesium Carbonate, Calcium Carbonate, Stevia Leaf Extract, Beet Powder Color, Safflower Oil. Nuun electrolytes contains (per tablet) the following: 3 grams of carbohydrate, calcium (15 mg, 1%DV), sodium (200 mg, 9%DV), potassium (125mg, 3%DV), magnesium (15mg, 4%DV), and chloride (75mg, 3%DV).

While Nuun Instant is commercially available and has received positive reviews from athletes, there have been no studies to date to evaluate the impact of this product or Nuun Electrolyte on hydration status. Therefore, the purpose of this study is to determine the impact of Nuun Instant powder and Nuun Electrolyte tablets on hydration status in young and active men and women. We will follow a similar approach as used by Maughan and colleagues (2016) to measure the fluid balance (the difference between the amount of water consumed and passed as urine) and beverage hydration index (the relative amount of urine passed after consumption of a drink compared to water), while also measuring plasma volume using the method of Dill and Costill (1974).

ELIGIBILITY:
Inclusion Criteria:

* body mass index (BMI) between 18-29.9 kg/m2
* no consumption of alcohol-containing beverages within 48 hours of testing
* no consumption of caffeine-containing beverages within 48 hours of testing
* no strenuous exercise within 48 hours of testing
* regularly consumes 2 liters of water daily
* engaged in structured exercise 3 or more hours per week for the past 6 months or longer

Exclusion Criteria:

* tobacco user
* active infection or illness
* pregnant

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-02-23 (Actual); Primary Completion 2021-04-06 (Actual); Study Completion 2021-04-06 (Actual)

PRIMARY OUTCOMES:
Body weight | baseline
  Body weight will be measured in underwear and papergown on digital scale.
Body weight | 4 hours after intervention
  Body weight will be measured in underwear and papergown on digital scale.
Urine Volume | Immediately following intervention
  Volume of urine output will be measured.
Urine Volume | 1 hour after intervention
  Volume of urine output will be measured.
Urine Volume | 2 hours after intervention
  Volume of urine output will be measured.
Urine Volume | 3 hours after intervention
  Volume of urine output will be measured.
Urine Volume | 4 hours after intervention
  Volume of urine output will be measured.
Urine Mass | immediately after intervention
  Urine output will be measured using an analytical scale.
Urine Mass | 1 hour after intervention
  Urine output will be measured using an analytical scale.
Urine Mass | 2 hours after intervention
  Urine output will be measured using an analytical scale.
Urine Mass | 3 hours after intervention
  Urine output will be measured using an analytical scale.
Urine Mass | 4 hours after intervention
  Urine output will be measured using an analytical scale.
Blood Pressure | baseline
  Blood Pressure will be measured.
Blood Pressure | 1 hour after intervention
  Blood Pressure will be measured.
Blood Pressure | 2 hours after intervention
  Blood Pressure will be measured.
Blood Pressure | 3 hours after intervention
  Blood Pressure will be measured.
Blood Pressure | 4 hours after intervention
  Blood Pressure will be measured.
Heart Rate | immediately after intervention
  Heart rate will be measured.
Heart Rate | 1 hour after intervention
  Heart rate will be measured.
Heart Rate | 2 hours after intervention
  Heart rate will be measured.
Heart Rate | 3 hours after intervention
  Heart rate will be measured.
Heart Rate | 4 hours after intervention
  Heart rate will be measured.
Hematocrit | baseline
  Hematocrit will be measured from blood.
Hematocrit | 4 hours after intervention
  Hematocrit will be measured from blood.
Hemoglobin | baseline
  Hemoglobin will be measured from blood.
Hemoglobin | 4 hours after intervention
  Hemoglobin will be measured from blood.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Bloomer, PhD, Principal Investigator — University of Memphis
Locations (1):
- Center for Nutraceutical and Dietary Supplement Reseach, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No